CLINICAL TRIAL: NCT01217203
Title: Multicenter Phase I Study on the Safety, Anti-tumor Activity and Pharmacology of IPH2101, a Human Monoclonal Anti-KIR, Combined With Lenalidomide in Patients With Multiple Myeloma Experiencing a First or Second Relapse
Brief Title: Study on the Safety, Anti-tumor Activity and Pharmacology of IPH2101 Combined With Lenalidomide in Patients With Multiple Myeloma Experiencing a First or Second Relapse
Acronym: KIRIMID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH2101-202
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Patients With Multiple Myeloma Experiencing a; First or Second Relapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPH2101 and lenalinomide (Experimental)
  Interventions: Drug: IPH2101 combined to lenalidomide

INTERVENTIONS:
Drug: IPH2101 combined to lenalidomide — Dose level 1 : 0.2 mg/kg IPH2101(with Lenalidomide 10 mg/day) Dose level 2 : 0.2 mg/kg IPH2101(with Lenalidomide 25 mg/day) Dose level 3 : 1 mg/kg IPH2101(with Lenalidomide 25 mg/day) Dose level 4 : 2 mg/kg IPH2101(with Lenalidomide 25 mg/day)
  Extension cohort: 6 patients at the Maximum Tolerated Dose (MTD)

SUMMARY:
The primary objective of the clinical study is to evaluate, in patients who experience a first or second relapse of their multiple myeloma, the safety of escalating doses of IPH2101 combined with lenalidomide

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any trial-related activities
2. Progressive disease or relapse of multiple myeloma (according to the IMWG definition) after one or two prior therapeutic treatments or regimens for multiple myeloma that achieved a response duration of at least 6 months
3. Prior therapeutic treatment regimens may have included Thalidomide and Lenalidomide. Regarding patients previously treated by Lenalidomide, only patients who achieved at least Partial Response duration of at least 6 months can be included. The patient must not have discontinued treatment due to Lenalidomide intolerance.
4. Measurable disease, as indicated by one or more of the following:

   * Serum M-protein ≥ 0.5 g/dL If Serum Protein Electrophoresis is felt to be unreliable for routine M-protein measurement (particularly for patients with IgA MM), then quantitative immunoglobulin levels can be accepted).
   * Urine Bence-Jones protein ≥ 200 mg/24 h
   * Involved serum Free Light Chains (sFLC) level ≥ 10 mg/dl ( ≥ 100 mg/l) provided sFLC ratio is abnormal (<0.26 or >1.65)
5. ECOG performance status of 0, 1 or 2
6. Clinical laboratory values at screening

   * Calculated creatinine clearance (according to MDRD) > 60 ml/min
   * Platelet ≥ 75 x 109 /l for patients with < 50% BM plasma cells, and ≥ 30 x 109 /l for patients with > 50% BM plasma cells
   * ANC > 1 x 109 /l
   * Bilirubin levels < 1.5 ULN ; ALT and AST < 3 ULN (grade 1 NCI)
7. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing Lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking Lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
8. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

1. Age < 18 years or > 80 years
2. Non secreting multiple myeloma or non measurable disease (< 0.5 g /dL M-Protein in serum or < 200 mg urinary M-protein / 24 h or <10 mg/dl involved sFLC)
3. Life-threatening conditions related or not to MM relapse
4. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking Lenalidomide)
5. Known hypersensitivity to thalidomide or IMiD®.
6. Use of any investigational agent within the last month
7. Treatment by systemic corticosteroids (except inhaled corticosteroids) or chemotherapy (including consolidation and maintenance) within the last month (use of biphosphonates is permitted)
8. Radiotherapy within the last month
9. Primary or associated amyloidosis
10. Peripheral neuropathy of grade ≥ 3 according to the CTCAE of the NCI
11. Abnormal cardiac status with any of the following

    * NYHA stage III or IV congestive heart failure
    * myocardial infarction within the previous 6 months
    * cardiac arrhythmia remaining symptomatic despite treatment
12. Current active infectious disease or positive serology for HIV, HCV or positive Hbs Antigen
13. History of or current auto-immune disease
14. History of other active malignancy within the past 5 years (apart from basal cell carcinoma of the skin, or in situ cervix carcinoma)
15. Serious concurrent uncontrolled medical disorder
16. History of allograft or solid organ transplantation
17. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
18. Inability to comply with an antithrombotic regimen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
number of patients with Dose Limiting Toxicity (DLT) at each dose level | 1 year
  safety of IPH2101 combined with lenalidomide at different dose levels.

SECONDARY OUTCOMES:
To assess response rate of the combination | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Don Benson, MD, Principal Investigator — The Ohio State University Comprehensive Cancer Center - Columbus OH - USA
Locations (6):
- United States (6):
  - Dana Farber, Boston, Massachusetts
  - NYU Clinical Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Saint Francis Hospital, Greensville, South Carolina

REFERENCES:
- [Derived] Benson DM Jr, Cohen AD, Jagannath S, Munshi NC, Spitzer G, Hofmeister CC, Efebera YA, Andre P, Zerbib R, Caligiuri MA. A Phase I Trial of the Anti-KIR Antibody IPH2101 and Lenalidomide in Patients with Relapsed/Refractory Multiple Myeloma. Clin Cancer Res. 2015 Sep 15;21(18):4055-61. doi: 10.1158/1078-0432.CCR-15-0304. Epub 2015 May 21. PMID 25999435